CLINICAL TRIAL: NCT04442906
Title: Comparative Study Between Dexmedetomidine and Fentanyl as an Adjuvant to Intra-articular Bupivacaine for Postoperative Analgesia After Knee Arthroscopy.
Brief Title: Analgesia After Knee Arthroscopy :Dexmedetomidine vs Fentanyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, Principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5355
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Analgesia
Keywords: dexmedetomidine; fentanyl; bupivacaine; knee arthroscopy; postoperative analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Fentanyl; Bupivacaine

STUDY DESIGN:
Intervention Model Description: analgesia for postoperative pain after knee arthroscopy: dexmedetomidine+bupivacaine, fentanyl+bupivacaine , bupivacaine
Who Masked: Participant, Outcomes Assessor
Masking Description: anesthetist not sharing in the study will assess patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group B (Active Comparator): IGroup B received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 ml saline
  Interventions: Drug: Bupivacain
- group BD (Active Comparator): . Group BD received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 ml dexmedetomidine (100 ug).
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacain
- group BF (Active Comparator): Group BF received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 fentanyl (50 ug).
  Interventions: Drug: Fentanyl; Drug: Bupivacain

INTERVENTIONS:
Drug: Dexmedetomidine — Group BD received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 ml dexmedetomidine (100 ug).
  Other Names: precedex
  Arms: group BD
Drug: Fentanyl — Group BF received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 fentanyl (50 ug)
  Arms: group BF
Drug: Bupivacain — Group B received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 ml saline.
  Other Names: marcaine

SUMMARY:
The aim of this study is to evaluate analgesic effects Bupivacaine, Bupivacaine plus Dexmedetomidine and Bupivacaine plus Fentanyl in relieving pain after knee arthroscopic surgery.

DETAILED DESCRIPTION:
Forty-five patients ASA I - II aged 21-45 years for elective knee arthroscopy were divided into 3 groups: Group B, BD and BF. Group B received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 ml saline. Group BD received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 ml dexmedetomidine (100 ug).

Group BF received Intra-articular injection of 20 ml bupivacaine 0.25%+ 1 fentanyl (50 ug). The time of first request of analgesia and analgesic effect by VAS during the first 24 hr. postoperatively are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Either sex,
* Age 21-45 years,
* American Society of Anesthesia (ASA) I - II for elective knee arthroscopy.

Exclusion Criteria:

* The patients with history of hepatic and renal diseases, psychiatric disorders,
* Prolonged intake of (NSAIDS, opioids and tricyclic antidepressant),
* Allergy to study drugs and patient who received analgesics up to 24 hr. before surgery were excluded from this study.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | For 24 hours postoperative
  start from intra-articular injection of the drug to the time of first request of analgesia

SECONDARY OUTCOMES:
total dose of rescue analgesia ( pethidine) | within 24 hours postoperative
  total consumption of rescue analgesia (pethidine) postoperative
The number of participants with bradycardia, itching and hypotension | Within 24 hours postoperative
  The number of participants with bradycardia less than 50 beat per minute, itching and hypotension if mean arterial blood pressure less than 20% of basal )
patient satisfaction | within 24 hours postoperative
  Patient satisfaction by five point Likert-Like verbal rating scale by asking the patient how they evaluate the experience with the analgesic management after the the surgery? (5-very satisfied, 4-satisfied, 3-neutral, 2-dissatisfied, 1-very dissatisfied)
pain intensity at rest (static) | measured immediately preoperative 0 minute ( admission receiving area)
  measured by VAS on 0-10 cm scale (0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 30 minutes postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 1 hour postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 2 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 4 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 6 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 8 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 12 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 18 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity at rest (static) | at 24 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | measured immediately preoperative 0 minute ( admission receiving area)
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 30 minutes postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 1 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 2 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 4 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 6 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 8 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 12 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 18 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)
pain intensity on mobilization of operated knee (dynamic) | at 24 hours postoperative
  measured by VAS on 0-10 cm scale(0- no pain and 10-the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Salem, MD., Principal Investigator — faculty of medicine , Zagazig University
Locations (1):
- Zagazig university, Zagazig, Egypt

REFERENCES:
- [Derived] Salem DAE, Nabi SMA, Alagamy SA, Kamel AAF. Comparative Study Between Dexmedetomidine and Fentanyl as an Adjuvant to Intraarticular Bupivacaine for Postoperative Analgesia after Knee Arthroscopy. Pain Physician. 2021 Nov;24(7):E989-E996. PMID 34704709